CLINICAL TRIAL: NCT07091916
Title: ExtraVascular Implantable Cardioverter Defibrillator (EV ICD) Japan Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MDT22010
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Tachycardia; Ventricular Arrythmia
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Implant Attempt (Experimental): Patients will be implanted with an extravascular ICD and undergo requisite electrical testing.
  Interventions: Device: Defibrillation using the Extravascular ICD

INTERVENTIONS:
Device: Defibrillation using the Extravascular ICD — VT/VF induction attempted for defibrillation testing, as well as requisite electrical testing.

SUMMARY:
The study is designed to characterize the acute safety and performance of the EV ICD System for Japanese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a Class I or IIa indication for implantation of an ICD according to the ACC/AHA/HRS Guidelines [i], or ESC guidelines [ii].
* Patient is at least 18 years of age and meets age requirements per local law.
* Patient is geographically stable and willing and able to complete the study procedures and visits for the duration of the follow-up.

  [i] Al-Khatib SM, Stevenson WG, Ackerman MJ, Bryant WJ, Callans DJ, Curtis AB, Deal BJ, Dickfeld T, Field ME, Fonarow GC, Gillis AM, Hlatky MA, Granger CB, Hammill SC, Joglar JA, Kay GN, Matlock DD, Myerburg RJ, Page RL. 2017 AHA/ACC/HRS guideline for management of patients with ventricular arrhythmias. [ii] Priori SG, Blomstrom-Lundqvist C, Mazzanti A, Blom N, Borggrefe M, Camm J, Elliot PM, Fitzsimons D, Hatala R, Hindricks G, Kirchhof P, Kjeldsen K, Kuck KH, Hernandez-Madrid A, Nikolaou N, Norekval TM, Spaulding C, Van Veldhuisen DJ. 2015 ESC guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death. European Heart Journal 2015 36:41 (2793-2867). https://doi.org/10.1093/eurheartj/ehv316

Exclusion Criteria:

* Patient is unwilling or unable to personally provide Informed Consent.
* Patient has indications for bradycardia pacing [iii] or Cardiac Resynchronization Therapy (CRT) [iv] (Class I, IIa, or IIb indication).
* Patient with an existing pacemaker, ICD, or CRT device implant or leads.
* Patients with these medical interventions are excluded from participation in the study:

  * Prior sternotomy
  * Any prior medical condition or procedure that leads to adhesions in the anterior mediastinal space (i.e., prior mediastinal instrumentation, mediastinitis)
  * Prior abdominal surgery in the epigastric region
  * Planned sternotomy
  * Prior chest radiotherapy

Or any other prior/planned medical intervention not listed that precludes their participation in the opinion of the Investigator.

* Patient has previous pericarditis that:

  * Was chronic and recurrent, or
  * Resulted in pericardial effusion [v], or
  * Resulted in pericardial thickening or calcification [vi].
* Patients with these medical conditions or anatomies are excluded from participation in the study:

  * Hiatal hernia that distorts mediastinal anatomy
  * Marked sternal abnormality (e.g., pectus excavatum)
  * Decompensated heart failure
  * COPD with oxygen dependence
  * Gross hepatosplenomegaly Or any other known medical condition or anatomy type not listed that precludes their participation in the opinion of the Investigator.
* Patients with a medical condition that precludes them from undergoing defibrillation testing:

  * Severe aortic stenosis
  * Intracardiac LA or LV thrombus
  * Severe proximal three-vessel or left main coronary artery disease without revascularization
  * Hemodynamic instability
  * Unstable angina
  * Recent stroke or transient ischemic attack (within the last 6 months)
  * Known inadequate external defibrillation
  * LVEF <20%
  * LVEDD >70 mm Or any other known medical condition not listed that precludes their participation in the opinion of the Investigator.
* Patient with any evidence of active infection or undergoing treatment for an infection.
* Patient is contraindicated from temporary suspension of oral/systemic anticoagulation
* Patient with current implantation of neurostimulator or any other chronically implanted device that delivers current in the body.
* Patient meets ACC/AHA/HRS or ESC clinical guideline Class III criteria for an ICD (e.g., life expectancy of less than 12 months).
* Patient is enrolled or planning to enroll in a concurrent clinical study that may confound the results of this study, without documented pre-approval from a Medtronic study manager.
* Patient with any exclusion criteria as required by local law (e.g., age or other).
* Pregnant women or breastfeeding women, or women of child bearing potential and who are not on a reliable form of birth regulation method or abstinence.

[iii] 2015 HRS/EHRA/APHRS/SOLAECE expert consensus statement on optimal implantable cardioverter-defibrillator programming and testing). [iv] ACC/AHA/HRS guidelines for Cardiac Resynchronization Therapy. [v] As documented on echo or MRI. [vi] As documented on CT scan or MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2025-01-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medtronic Japan Co., Ltd., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first site was activated on 20JAN2023. The first EV ICD Japan subject was enrolled on 22FEB2023 and implanted on 01 MAR 2023. The last subject enrollment occurred on 27SEP2023, and the last implant occurred on 03OCT2023. Sites were notified of enrollment completion on 01DEC2023.
Groups:
- Implant Attempt: Subjects undergoing an implant attempt of an Extravascular ICD System, including implant testing (sensing, impedance and pacing testing) and induction and defibrillation testing using the Extravascular ICD.
Period: Overall Study
Arm/Group | Implant Attempt
Started (Subjects who underwent an implant attempt of the Extravascular ICD System) | 14
Completed (Subjects followed up at least to the 2-week visit after the Extravascular ICD System having been fully implanted) | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects who underwent an implant attempt of the Extravascular ICD System
Groups:
- Implant Attempt EV ICD Japan: Subjects undergoing an implant attempt of an Extravascular ICD System, including implant testing (sensing, impedance and pacing testing) and induction and defibrillation testing using the Extravascular ICD.
Arm/Group | Implant Attempt EV ICD Japan
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety Outcome - Freedom From Major Complications Related to the EV ICD System and/or Procedure at 2 Weeks Post-implant
Description: The endpoint is defined as a subject's first occurrence of a major complication related to the EV ICD System and/or procedure, as determined by an independent Clinical Events Committee (CEC), that occurs on or prior to 2 weeks (14 days) post-implant.
Time Frame: 2 weeks (14 days) post-implant
Measure: Count of Participants; unit: Participants
Arm/Group | Implant Attempt
Number analyzed (Participants) | 14
Participants | 13
Statistical Analysis 1: Comparison: Implant Attempt; The first primary objective is to characterize the freedom from major complications related to the EV ICD System and/or procedure at 2 weeks post-implant. The endpoint is defined as a subject's first occurrence of a major complication related to the EV ICD System and/or procedure, as determined by an independent Clinical Events Committee (CEC), that occurs on or prior to 2 weeks (14 days) post-implant; Test type: Other — This objective was for the purpose of gathering data pertaining to device safety over the first 2 weeks post-implant. There were no pre-specified performance criteria or hypotheses for this objective; descriptive statistics; Proportion = 92.9

2. Primary Outcome: Efficacy Outcome - Defibrillation Efficacy at Implant of the EV ICD System
Description: Each subject will demonstrate a successful defibrillation outcome if either 2 successive induced ventricular fibrillation episodes are terminated by the subject's device delivering a shock at the required energy level, or if one such episode is successfully terminated by the subject's device delivering a shock at a lower energy level. Up to 6 such episodes may be induced to test device efficacy.
Time Frame: At Implant
Measure: Count of Participants; unit: Participants
Arm/Group | Implant Attempt
Number analyzed (Participants) | 14
Participants | 14
Statistical Analysis 1: Comparison: Implant Attempt; The primary efficacy objective was to characterize the defibrillation efficacy at implant of the EV ICD System; Test type: Other — There were no hypotheses for this objective; descriptive statistics; Proportion = 100

ADVERSE EVENTS:
Time Frame: Among the 14 enrolled subjects, the average follow-up duration from enrollment to last documented contact was 112.9 ± 59.9 days.
Description: All adverse events (AEs) are collected throughout the study duration, starting at the time the Informed Consent Form is signed.
  Reporting of these events to Medtronic will occur on an Adverse Event eCRF, including a description of AE, date of onset of AE, date of awareness of site, treatment, resolution, assessment of both the seriousness and the relatedness to the system and/or procedure.
  The Pivotal Study used MedDRA 26.0
Groups:
- Enrolled Japan Study: Subjects enrolled in the Extravascular ICD Japan Study
Arm/Group | Enrolled Japan Study
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 5/14
Other Adverse Events (participants affected / at risk) | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Japan Study (N=14)
Incision site pain (Injury, poisoning and procedural complications) | 3 (3)
Cardiac perforation (Cardiac disorders) | 1 (1)
Device inversion (Product Issues) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Japan Study (N=14)
Inflammation (General disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic gastritis (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Medical device site pain (General disorders) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Renal cyst infection (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Device pacing issue (Product Issues) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT07091916/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT07091916/SAP_001.pdf